CLINICAL TRIAL: NCT03156920
Title: Pretreatment With Sumatriptan on Cilostazol Induced Headache in Healthy Volunteers. Development of a Pragmatic Migraine Model
Brief Title: Pretreatment With Sumatriptan on Cilostazol Induced Headache in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Katrine Falkenberg, Medical doctor, PhD student, principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-15011960
Record Dates: First submitted 2017-05-10; First posted 2017-05-17 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sumatriptan (Active Comparator): Headache is induced with Cilostazol. This headache is pre-treated double-blinded with 2 tablets of sumatriptan 50 mg
  Interventions: Drug: Sumatriptan
- Placebo (Placebo Comparator): Headache is induced with Cilostazol. This headache is pre-treated double-blinded with 2 tablets of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Cilostazol is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Arms: Placebo
Drug: Sumatriptan — Cilostazol is given both study days to induce headache. One day the headache is treated with placebo and the other day with sumatriptan
  Arms: Sumatriptan

SUMMARY:
To develop a pragmatic migraine model the investigators will induce headache in healthy volunteers with a phosphodiesterase inhibitor (cilostazol). The participants will be pre-treated with sumatriptan. If the headache responds to sumatriptan, the model can be used to test new drug candidates.

DETAILED DESCRIPTION:
There remains a great need for more effective anti-migraine drugs with fewer side effects. Human experimental models are valuable in early phase development of new anti-migraine drugs but useful models have not yet been developed. The investigators' group has shown that Cilostazol, a phosphodiesterase inhibitor induce headache/migraine in both healthy volunteers and in patients with migraine without aura (MO).

To validate cilostazol as a model, the headache must respond to specific migraine treatment with sumatriptan.

Hypothesis: Cilostazol induces a migraine-like headache in healthy subjects. The induced headache can be pre-treated with a specific anti-migraine drug; sumatriptan.

Aim: Developing a pragmatic and valid model for the testing of new anti-migraine drugs.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects of both sexes Age 18-60 years Weight 50-95 kg. Females were requested to use effective contraception.

Exclusion Criteria:

Any type of headache (except episodic tension-type headache < 1 day per week) Serious somatic or psychiatric disease Pregnancy Intake of daily medication (except oral contraceptives).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Difference in median headache score 2 hours after cilostazol | 2 hours
  The investigators will assess the outcome measures 1 year after the beginning of the study
Area under the headache score curve | 12 hours
  The investigators will assess the outcome measures 1 year after the beginning of the study

SECONDARY OUTCOMES:
Difference in peak headache score | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Katrine Falkenberg, Copenhagen, Glostrup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falkenberg K, Olesen J. Pre-treatment with sumatriptan for cilostazol induced headache in healthy volunteers. J Headache Pain. 2018 Aug 17;19(1):71. doi: 10.1186/s10194-018-0890-y. PMID 30120600